CLINICAL TRIAL: NCT03029533
Title: An Open Label, Randomized, Single Dose, Parallel-group, Phase 1 Study to Evaluate the Pharmacokinetics and Safety Following Subcutaneous Administration of DWJ108J in Patients With Prostate Cancer
Brief Title: Phase 1 Study to Evaluate the Pharmacokinetics and Safety Following SC Administration of DWJ108J in Patients With Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_LP3M002
Record Dates: First submitted 2017-01-12; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DWJ108J (leuprolide acetate) (Experimental): DWJ108J (leuprolide acetate)
  Interventions: Drug: Leuprolide Acetate
- Leuplin DPS Inj (Active Comparator): Leuplin DPS Inj
  Interventions: Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Leuprolide Acetate — DWJ108J, SC injection, once(Day1)
  Other Names: DWJ108J
  Arms: DWJ108J (leuprolide acetate)
Drug: Leuprolide Acetate — Leuplin DPS Inj, SC injection, once(Day1)
  Other Names: Leuplin DPS Inj
  Arms: Leuplin DPS Inj

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety of DWJ108J (leuprolide acetate) and Leuplin DPS Inj administered subcutaneously in patients with prostate cancer

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥19 and ≤80 years of age at Screening.
2. Subject with histologically proven adenocarcinoma of the prostate requiring androgen deprivation therapy
3. An ECOG performance status grade of 0 to 2,
4. 19kg/m2≤ Body Mass Index (BMI) ≤30kg/m2 at Screening.

Exclusion Criteria:

1. Confirmed Hormone refractory prostate cancer(HRPC)
2. Has had history of bilateral orchiectomy, suprarenalectomy or hypophysectomy.
3. Diagnosed pituitary adenoma
4. Has a history of depression
5. Has a risk of spinal cor d compression due to metastatic spinal cord injury.
6. Has a severe urethratresia.
7. Confirmed uncontrolled Congestive heart failure (CHF) within 6 months of Screening.
8. Has a history of MI or any procedure with regard to coronary artery disease within 6 months of Screening. (e.g., balloon angioplasty, coronary artery bypass graft)
9. Has any severe concomitant disease that would interfere with the conduct of the study except for prostate cancer
10. Has allergy history of leuprolide acetate, similar GnRH drugs or other medications (e.g., Aspirin, antibiotics) and/or has any allergic disease requiring treatment.
11. Has received an investigational drug within 9 0days of Screening.
12. Drug releasing is expected after administration of study drug, if subject received GnRH agonist for treatment of prostate cancer.
13. Has other chemotherapy planned within 14weeks from administration of study drug, except for androgen deprivation therapy.
14. Has no willing of using method of contraception throughout the study period.
15. Systolic Blood Pressure < 90mmHg and/or ≥160mmHg or Diastolic Blood Pressure < 60mmHg and/or ≥100mmHg at Screening
16. QTcF >450msec at Screening ECG.
17. HbA1c level is high the upper limit of normal of reference range.
18. Serum AST, ALT or Creatinine > 1.5times the upper limit of normal at Screening.
19. Positive results of tests for hepatitis B, hepatitis C, HIV or syphilis.
20. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest of the subject.

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day 99
Area under the plasma concentration versus time curve (AUC) | Day 99
  AUC0-7, AUC7-28, AUC 0-42, AUCt, AUCinf